CLINICAL TRIAL: NCT02250287
Title: Pilot and Feasibility Study: Evaluation of New Quantitative Magnetic Resonance Imaging Parameters in Assessing the Kidneys of Autosomal Dominant Polycystic Kidney Disease
Brief Title: New Quantitive MRI Parameters in Assessing Kidneys of Autosomal Dominant Polycystic Kidney Disease
Acronym: MRI Pilot
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Sudhakar K. Venkatesh, M.D., Primary Investigator, Mayo Clinic
Other Study IDs: 14-000866
Record Dates: First submitted 2014-09-18; First posted 2014-09-26 (Estimated); Last update posted 2016-06-17 (Estimated); Status verified 2016-05

CONDITIONS: Autosomal Dominant Polycystic Kidney Disease; Kidney Disease
Keywords: autosomal dominant polycystic kidney disease; magnetic resonance imaging parameters; magnetic resonance elastography; apparent diffusion coefficient; blood oxygen level determinations; diffusion weighted imaging
MeSH Terms: conditions — Polycystic Kidney, Autosomal Dominant; Kidney Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to establish normal Magnetic Resonance quantitative values (tissues stiffness, Apparent Diffusion Coefficient values and Blood Oxygen Level Determination values for both renal cortex and medullary tissues and total renal blood flow) for young Autosomal Dominant Polycystic Kidney Disease patients with normal renal function, and normal young adult controls without Autosomal Dominant Polycystic Kidney Disease and normal renal function.

Hypothesis: Newer Magnetic Resonance quantitative imaging parameters (tissue stiffness, Apparent Diffusion Coefficient, Blood Oxygen Level Determination levels, Magnetization Transfer and renal blood flow) will have different values in young adult ADPKD patients as compared to normal volunteers.

ELIGIBILITY:
Inclusion criteria ADPKD participants

* Male and female subjects between 18-30 years of age
* Diagnosis of ADPKD
* Glomerular Filtration Rate (GFR) of > or = to 60 mL/min (Chronic Kidney Disease-Epidemiology Collaboration equation)
* Ability to provide written, informed consent

Exclusion criteria for ADPKD participants

* Clinically significant concomitant systemic disease
* Subjects with Diabetes Mellitus
* Urinary protein excretion
* Abnormal urinalysis suggestive of concomitant glomerular disease
* Subjects having contraindications to, or interference with MRI assessments
* Subjects with supine blood pressure higher than 140/90 mm Hg or taking blood pressure medications

Inclusion criteria for Normal Volunteers

* Male and female subjects between 18-30 years of age
* Glomerular Filtration Rate (GFR) of > or = to 60 mL/min (Chronic Kidney Disease-Epidemiology Collaboration equation)
* Ability to provide written, informed consent

Exclusion criteria for Normal Volunteers

* Previous personal or family history of kidney disease
* Clinically significant concomitant systemic disease
* Subjects with Diabetes Mellitus
* Urinary protein excretion
* Abnormal urinalysis suggestive of concomitant glomerular disease
* Subjects having contraindications to, or interference with MRI assessments
* Subjects with supine blood pressure higher than 140/90 mm Hg or taking blood pressure medications

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Ten known ADPKD patients between the ages of 18-30, and 10 normal non-ADPKD volunteers between the ages of 18-30, who are MRI compatible will be studied. Study participants will be selected from a list queried from the Polycystic Kidney Disease database.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2014-12; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Evaluate renal tissue stiffness | baseline
  The renal parenchymal tissue stiffness is measured in kilopascals with magnetic resonance elastography sequence.
Magnetization transfer ratio | baseline
  The magnetization transfer ratio of renal tissue is measured with magnetization transfer sequence and expressed as a ratio.
Diffusion | baseline
  Diffusion is quantified as apparent diffusion coefficient (x10-3/mm2) in renal tissue is measured with intravoxel incoherent motion imaging (IVIM) sequence and diffusion tensor imaging (DTI).
Perfusion quantified as blood flow in mL/s. | baseline
  Perfusion in the renal tissue is measured with arterial spin labeling sequence and phase contrast magnetic resonance angiography.

CONTACTS AND LOCATIONS:
Overall Officials: Sudhakar Venkatesh, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States